CLINICAL TRIAL: NCT00980577
Title: Phase 2 Study of Stimulating Catheter for Continuous Femoral Nerve Block in Total Knee Replacement
Brief Title: Stimulating Catheter With or Without Ultrasound Guidance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Peng Ruicong, Peking University Health Science Center Review Board
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PUTH7275
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2009-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NS (Active Comparator): stimulating catheter will be inserted using stimulator
  Interventions: Device: NUUS

INTERVENTIONS:
Device: NUUS — Sonosite Micro Maxx
  Other Names: stimulating catheter will be inserted under stimulator and ungrasoud guidance

SUMMARY:
To study whether the combination of ultrasound guidance and stimulating catheter could reduce the time for needle and catheter insertion compared with using stimulating catheter alone. Secondary outcomes: analgesic effects after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective primary total knee replacement surgery under neuraxial anesthesia ASA<=4
* Able to give informed consent
* Able to cooperate with sensory and motor testing of lower limb function

Exclusion Criteria:

* coagulopathy
* Allergy to local anaesthetic or postanalgesic rescue regimen
* Signs, symptoms or laboratory evidence of local infection or systemic sepsis
* No pre-existing neurological deficit (sensory or motor) affecting lower limb
* Patients with lower limb amputations

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
time and number of attempts to perform block, the efficacy of the block | during the block procedure

SECONDARY OUTCOMES:
postoperative analgesic effect | pod 1-3

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hosptial, Beijing, China